CLINICAL TRIAL: NCT05436795
Title: Evaluation of the Impact of a Digital Self-testing Strategy in Individuals With Suspected COVID-19 Infection in South Africa on Time to Action Plans, Linkage to Care, Detection of New Infections: A Randomized Controlled Superiority Trial.
Brief Title: A Randomized Controlled Trial of a Digital, Self-testing Strategy for COVID-19 Infection in South Africa.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: University of Cape Town Lung Institute (Other)
Responsible Party: Principal Investigator, Nitika Pai, Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 174921
Record Dates: First submitted 2022-06-27; First posted 2022-06-29 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: COVID-19
Keywords: COVID-19; self-test; self-sample; point-of-care; randomized controlled trial; rapid test; digital; app-based; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome evaluator (statistician) will be unaware of the intervention allocation (single-blind).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Arm (Experimental): In the interventional arm, we will offer a self-administered supervised COVID-19 testing strategy with an investigational device - Abbott's Panbio COVID-19 Antigen Self-test. The self-test process will be facilitated by the COVIDSmart CARE! digital App and platform. Suspected COVID-19 patients will be triaged into one of three action plans: a) clinical care pathways, b) prevention (home quarantine, isolation) pathways, or c) social distancing.
  Interventions: Device: Abbott Panbio rapid antigen self-tests; Other: COVIDSmart CARE! app
- Conventional Arm (No Intervention): Participants presenting to test for SARS-CoV-2 will be staged on their self-reported severity of symptoms (mild, moderate, severe) and tested with rapid antigen tests, followed by RT-PCR testing. Suspected COVID-19 patients will be triaged into one of three action plans: a) clinical care pathways, b) prevention (home quarantine, isolation) pathways, or c) social distancing.
  Conventional arm is the standard of care arm.

INTERVENTIONS:
Device: Abbott Panbio rapid antigen self-tests — COVID-19 self-testing will be performed using investigational Abbott Panbio rapid antigen self-test kits that require self-sampled nasal swabs.
  Arms: Interventional Arm
Other: COVIDSmart CARE! app — Guided by the application that connects, educates, and communicates a digital, contactless open access strategy, participants will have the opportunity to self-test and assess their risk level of COVID-19 infection, as well as the option to refer their close contacts to testing for those who are COVID-19 positive, through the study platform.
  Arms: Interventional Arm

SUMMARY:
As the world opens up to rapidly increasing vaccination coverage and newer variants, there is an even greater need for timely access to at-home COVID-19 testing, or self-testing based out of kiosks, offices, or private spaces.

Data on digital strategies that complement self-testing are sparse. Using a superiority randomized controlled trial design (open-label, single-blinded), the investigators will aim to evaluate the impact of a digital self-testing strategy offered out of kiosks/private spaces on the turnaround time to test results, the proportion of participants initiated on action plans, and new infection detected with the strategy. The investigators will compare these outcomes to a conventional lab-based strategy.

Significance:

A digital, portable, self-testing strategy will facilitate rapid self-knowledge of COVID-19 status and rapid classification into clinical/quarantine/prevention plans.

The study will document the impact of a digitally connected self-testing strategy for COVID-19 infection. Upon completion of the strategy, the digital program will be available for global dissemination.

DETAILED DESCRIPTION:
The investigators hypothesize that a rapid digital self-testing strategy that evaluates the risk of severe COVID-19 infection and guides participants on the methods of self-test interpretation and ensuing action plans will be more impactful in detecting COVID-19 infection and will facilitate more participants to take an appropriate course of action compared to the conventional strategy. Action plans initiated will be either: a) clinical care, b) prevention (home quarantine, isolation), or c) social distancing. Taken together, these actions will impact health outcomes during the current and ensuing SARS-CoV-2 surges.

Using a superiority randomized controlled trial (RCT) design, the investigators will randomize participants to either the App-based self-testing arm or the conventional testing arm (screening and testing performed by a health care worker (HCW) at the COVID-19 testing site). A confirmatory RT-PCR test will be performed in both arms. The standard of care will be offered in the conventional arm.

The interventional strategy will be offered in kiosks/private spaces within COVID-19 testing sites or student health clinics. The COVIDSmart CARE! digital App-based program will be downloaded onto the test kiosk based tablets or participants' smartphones. This strategy will yield self-test results and guided action plans in a rapid turnaround time.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above
* All sexes and genders
* Suspecting COVID-19 exposure
* Symptomatic or asymptomatic for COVID-19
* Mental capacity to provide informed consent
* Access to internet connectivity and digitally literate
* Access to a smart device that can download and run the COVIDSmart CARE! App (e.g., Android tablet version 6 or higher).

Exclusion Criteria:

* Participants with serious mental health or clinical condition which limits their capacity to provide informed consent.
* Those with apparent severe COVID-19 symptoms requiring urgent hospitalization (e.g., severe shortness of breath, impaired level of consciousness, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Estimating the impact on turnaround time (TAT) from the point of taking a test to initiating a clinical action plan. | Less than 24-48 hours
  TAT is estimated to be <2 hours compared to 24 hours taken with a conventional RT-PCR test.

SECONDARY OUTCOMES:
The impact of the COVIDSmart CARE! self-testing strategy on the proportion of participants taking an appropriate COVID-19 related action compared to conventional COVID-19 testing strategies at 24 hours post randomization. | Less than 24-48 hours
  Proportional estimates of participants who action the guidance given via the App compared to those who undergo standard of care testing will measure the efficacy of the App on changing behaviour and/or linkage to care.
Impact on detection of new COVID-19 infections in each arm. | 1 year
  We will document the impact of digital self-testing versus conventional testing on the number of new COVID-19 infections detected in each arm. We will compare and document the proportion of newly identified participants as test positives in both arms. Test positives and test negatives will be confirmed by lab confirmed results and test protocols.

OTHER OUTCOMES:
Diagnostic accuracy of COVIDSmart CARE! versus conventional reference standard. | 1 year
  We will compare the diagnostic performance of our interventional (digital self-testing strategy) versus conventional RT-PCR tested (a composite reference standard algorithm containing NAATs from a different manufacturer); with performance metrics (i.e., sensitivity, specificity, and positive and negative predictive values with 95% CI).

CONTACTS AND LOCATIONS:
Overall Officials: Nitika Pant Pai, MD, MPH, PhD, Principal Investigator — McGill University Health Centre Research Institute, Montreal, Canada
Locations (1):
- University of Cape Town Lung Institute, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No